CLINICAL TRIAL: NCT03443349
Title: A Single - Centre Safety Study About the Safety, Practicability and Acceptance of "Vibwife One", a New Medical Device to Support Delivering Women in Their Mobilization
Brief Title: "Vibwife One" a New Medical Device to Support Delivering Women in Their Mobilization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Clinical Trial Unit, University Hospital Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2017-02085
Record Dates: First submitted 2018-01-02; First posted 2018-02-23 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Medical Device
Keywords: Delivering Women

STUDY DESIGN:
Intervention Model Description: The medical device will be used according to its market authorization, i.e. CE-Certification. Because it will be used for the first time in pregnant women, a vulnerable population, the following three step application procedure has been determined:
  * First five pregnant women use the device for 10 minutes. Each of them in a position and module proposed by the midwife with the agreement of the woman.
  * Next 10 pregnant women use the device for 20 minutes. Again, position and module according to the decision of the midwife in agreement with the woman.
  * All the remaining pregnant women (35) use the device for 30 minutes. Position and module proposed by the midwife with the agreement of the woman.
  During the intervention period, position and module might be changed once if required.
  There will be a safety review board meeting after each group of the pregnant women having used the device, checking the safety criteria according to predefined Adverse Device Effects and Adverse Events.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Use of the medical Device: Vibwife One (Other): The medical device will be used according to its market authorization.
  Because it will be used for the first time in pregnant women, the following three step application procedure has been determined:
  * First five pregnant women use the device for 10 minutes. Each of them in a position and module proposed by the midwife with the agreement of the woman.
  * Next 10 pregnant women use the device for 20 minutes. Again, position and module according to the decision of the midwife with the agreement of the woman.
  * All the remaining pregnant women (35) use the device for 30 minutes. Position and module according to the decision of the midwife with the agreement of the woman.
  During the intervention period, position and module might be changed once if required.
  Interventions: Device: Vibwife One

INTERVENTIONS:
Device: Vibwife One — Vibwife One is a powered rotation bed intended to be used to assist in active mobilization of delivering women. "Vibwife One" imitates manual mobilization and position techniques. It is integrated in the mattress and fixed to the pelvis area of the birthing bed. "Vibwife One" can be used, when manual mobilization and position techniques are deemed appropriate.
  The device with all its functions is controlled over a remote control.

SUMMARY:
"Vibwife One" was developed to support the mobilization of the delivering women during the labor process. It consists of a mattress that fits on existing delivery beds. Different movements, adjustable in pace and intensity can be chosen to mobilize women in labor.

Although existing evidence is rare, some literature and historical reports have shown a positive impact of active mobilization during labor.

At time of rising epidural anesthesia rate, "Vibwife One" could be an interesting way to active mobilize those women to support the physiological birth process.

So far, the device has not yet been applied in delivering women. The investigators carry out a first safety study to assess the safety, to evaluate the comfort and the practicability for delivering women and medical staff of this new medical device.

DETAILED DESCRIPTION:
The medical device will be used according to its market authorization. Because it will be used for the first time in pregnant women, the following three step application procedure has been determined:

* First five pregnant women use the device for 10 minutes. Each of them in a position and module proposed by the midwife with the agreement of the woman.
* Next 10 pregnant women use the device for 20 minutes. Again, position and module according to the decision of the midwife with the agreement of the woman.
* All the remaining pregnant women (35) use the device for 30 minutes. Position and module according to the decision of the midwife with the agreement of the woman.

During the intervention period, position and module might be changed once if required.

After the inclusion of all the 50 participants, each position and module has to be tested.

There will be a safety review board consisting of one physician, one midwife and a clinical expert midwife meeting after each group of pregnant women having used the device, evaluating the safety criteria according to predefined Adverse Device Effects and Adverse Events.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent documented by signature
* German or English speaking
* Singleton healthy pregnancy
* Cephalic presentation
* ≥37th weeks of gestation
* 4cm - 9cm of dilatation
* Regular contractions
* Physiological cardiotocograph (CTG) 30 min pre-intervention
* Physiological blood pressure (111/66 - 139/89)

Exclusion Criteria:

* Multiple pregnancies
* Breech position
* Small for gestational age (<10. Percentile)
* Fetal congenital abnormalities
* Placenta praevia
* Fetal distress
* Heavy vaginal bleeding during birth
* Maternal weight ≥ 135 kg
* Preeclampsia or HELLP
* Diabetes I and II / Gestational diabetes insulin dependent
* Spinal and back disorder (herniated disk / scoliosis)
* Hypertension (≥140/90 mmHg)
* Hypotension (Basic blood pressure in the third trimester -20%, if not available: ≤ 110/65 mmHg)
* No signed informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2018-01-23 (Actual); Primary Completion 2018-11-06 (Actual); Study Completion 2018-11-06 (Actual)

PRIMARY OUTCOMES:
Safety measured by number of Adverse Events and Adverse Device Effects | During intervention and until 30min. after end of intervention
  The Primary outcome is safety of the pregnant woman and the child using "Vibwife One" in the first stage of Labor. It will be evaluated according to predefined Adverse Events and Adverse Device Effects.

SECONDARY OUTCOMES:
Pain intensity | VAS before, during and after end of the intervention, intervention lasting up to 30 min.
  Pain intensity is measured by a discrete Visual Analogue Scale (VAS) from 0-10, 0 indicating no pain until 10 indicating greatest pain
Preferences measured by questionnaire | within 30 minutes after end of the intervention, intervention lasting up to 30 min.
  Women's preferences regarding the medical device will be measured by a questionnaire with a 4-issue Likert scale; Likert scaling is a bipolar scaling method, measuring either positive or negative response to a statement. The responses in this study might be 1.Strongly disagree, 2.Disagree, 3.Agree 4. Strongly agree, answers ranging from 1 point (strongly disagree) to 4 points (strongly agree). Low amount of points represent a better outcome.
Practicability measured by questionnaire | from first birth in the study until last birth in the study (start of study until study completion an average of 1 year)
  Practicability of the medical device and views of the midwives and physicians will be assessed by a questionnaire with a 4-issue Likert scale; Likert scaling is a bipolar scaling method, measuring either positive or negative response to a statement. The responses in this study might be 1.Strongly disagree, 2.Disagree, 3.Agree 4. Strongly agree, answers ranging from 1 point (strongly disagree) to 4 points (strongly agree). Low amount of points represent a better outcome.

OTHER OUTCOMES:
Duration of first stage of labor measured by hours | assessed during birth
  The first stage is defined from 4cm till full dilatation (10cm) of the cervix
Duration of second stage of labor measured by hours | assessed during birth
  The second stage is defined as part of labor from the full dilatation of the Cervix until birth
Delivery Outcome measured by frequency of route of delivery | from first birth in the study until last birth in the study (start of study until study completion an average of 1 year)
  Frequencies and means of characteristics of delivery (spontaneous versus vaginal instrumental versus caesarian section)

CONTACTS AND LOCATIONS:
Overall Officials: Irene Hösli, Prof. Dr. MD, Principal Investigator — Chief Physician Departement of Obstetrics and Antenatal care
Locations (1):
- University Hospital Basel, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lawrence A, Lewis L, Hofmeyr GJ, Styles C. Maternal positions and mobility during first stage labour. Cochrane Database Syst Rev. 2013 Aug 20;(8):CD003934. doi: 10.1002/14651858.CD003934.pub3. PMID 23959763
- [Background] Nieuwenhuijze MJ, de Jonge A, Korstjens I, Bude L, Lagro-Janssen TL. Influence on birthing positions affects women's sense of control in second stage of labour. Midwifery. 2013 Nov;29(11):e107-14. doi: 10.1016/j.midw.2012.12.007. Epub 2013 Feb 15. PMID 23415350